CLINICAL TRIAL: NCT01043198
Title: Phenotypic Characterization and Array CGH Analysis in Patients With Syndromic Obesity of Unknown Etiology
Brief Title: Microarray Analysis in Syndromic Obesity
Acronym: REMOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2009/26
Record Dates: First submitted 2009-12-29; First posted 2010-01-06 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Mental Retardation; Syndromic Obesity
Keywords: CGH array technology; mental retardation; chromosomal abnormalities; syndromic obesity; obesity
MeSH Terms: conditions — Intellectual Disability; Chromosome Aberrations; Obesity | interventions — Restraint, Physical; Blood Specimen Collection; Biological Products; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Clinical examination and blood sampling for biological and genetic analysis — Clinical examination and precise description of the phenotype (questionnaire)
  * Standardized screening with :
  * radiological (hands, feet, spine ; and renal ultrasonography)
  * biological (hormonal, metabolic, and "basic" genetic investigations (karyotype, FISH 22q11.2, Fragile X, and other depending on the clinical data))

SUMMARY:
Comparative genomic hybridization (CGH) array technology has been used in numerous studies on mental retardation, and few chromosomal abnormalities have been identified in patients. Because chromosomal abnormalities have still been associated with obesity, we can expect that syndromic obesity is also associated with small deletions/duplications. Characterization of deleted or duplicated loci in these obese patients would mean that these loci include genes implicated in obesity. This will permit to propose new gene(s) involved in obesity. (In french: Caractérisation phénotypique et recherche de REManiements chromosomiques chez des patients présentant une OBésité syndromique de cause non identifiée : REMOB)

DETAILED DESCRIPTION:
With the introduction of array comparative genomic hybridization (CGH), genome-wide high resolution analysis for DNA copy number alterations became feasible. This technology has been principally used in patients with mental retardation. Depending on the eligibility criteria and resolution of the array, around 10 % of patients with mental retardation are found with cryptic chromosomal imbalance. This figure arises 20 % for patients with mental retardation and multiple congenital anomalies. Alteration of the lipid metabolism and/or regulation of satiety, obesity (except in presence of other "exogen" factors) can be considered as a developmental disorder. Also, different syndromes with obesity have been associated with chromosomal abnormalities, such as 1p36 deletion syndrome, 2q37 deletion syndrome, chromosome 14 maternal disomy … So we can expect that syndromic obesity is similarly associated with sub cryptic chromosomal abnormalities. Some "isolated" patients with obesity have been described with cryptic chromosomal imbalance found by array CGH, but no study has been realized in cohorts of patients selected for syndromic obesity.

Characterization of cryptic chromosomal anomaly(ies) in a patient will also be useful to precise the management and follow-up of the patient and to give the family an adapted genetic counselling.

We will define a cohort of patients with syndromic obesity and propose them to realize a first screening looking for the "common" aetiologies of syndromic obesity. If this screening is normal, array CGH will be realized. This analysis implies a blood sampling of 5 ml in patient and his parents.

Genes present at the deleted or duplicated loci characterized in the patients will be study to determine if some could be specifically implicated in the development of obesity. These same genes could be implicated in isolated obesity. Our study will be also useful to precise the aetiological screening of syndromic obesity, and determine the place of array-CGH.

ELIGIBILITY:
Inclusion Criteria:

* children (under 18 year-old)
* obesity (following IOTF definition)
* at least one criteria among :

  * mental retardation
  * facial dysmorphism
  * at least one major malformation (uro-genital, cardiac, skeletal, cerebral, ophthalmologic…)

Exclusion Criteria:

* common obesity
* obesity with an identified aetiology

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the prevalence of cryptic chromosomal imbalance in patients with syndromic obesity of unknown etiology. | 3 - 6 months

SECONDARY OUTCOMES:
prevalence of the main genetic aetiologies of syndromic obesity | 3 - 6 months
Characterization of the main features evocative of subcryptic chromosomal anomalies in this population | 3 - 6 months
Phenotypic description of some "new" syndromes with obesity | 3 - 6 months
candidate genes implicated in the development of obesity. | 3 - 6 months
Delineation of an aetiological screening protocol in patients with syndromic obesity | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange DELRUE, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (6):
- France (6):
  - Service de Génétique de médicale - Hopital des enfants - Pellegrin, Bordeaux
  - Centre de Génétique Hôpital d'Enfants CHU de Dijon, Dijon
  - Génétique Médicale HOPITAL DEBROUSSE HCL, Lyon
  - Département de Génétique Médicale Centre de référence anomalies du développement Centre de compétence maladies osseuses constitutionnelles Hôpital Arnaud de Villeneuve CHRU Montpellier, Montpellier
  - Département de Génétique Hôpital Robert DEBRE Centre de Référence Maladies Rares "Anomalies du Développement & Syndromes Malformatifs", Paris
  - Hopital des Enfants, CHU de Toulouse, Toulouse

REFERENCES:
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Ichihara S, Yamada Y. Genetic factors for human obesity. Cell Mol Life Sci. 2008 Apr;65(7-8):1086-98. doi: 10.1007/s00018-007-7453-8. PMID 18097636
- [Background] Delrue MA, Michaud JL. Fat chance: genetic syndromes with obesity. Clin Genet. 2004 Aug;66(2):83-93. doi: 10.1111/j.0009-9163.2004.00300.x. PMID 15253756
- [Background] Schoumans J, Ruivenkamp C, Holmberg E, Kyllerman M, Anderlid BM, Nordenskjold M. Detection of chromosomal imbalances in children with idiopathic mental retardation by array based comparative genomic hybridisation (array-CGH). J Med Genet. 2005 Sep;42(9):699-705. doi: 10.1136/jmg.2004.029637. PMID 16141005
- [Background] Fan YS, Jayakar P, Zhu H, Barbouth D, Sacharow S, Morales A, Carver V, Benke P, Mundy P, Elsas LJ. Detection of pathogenic gene copy number variations in patients with mental retardation by genomewide oligonucleotide array comparative genomic hybridization. Hum Mutat. 2007 Nov;28(11):1124-32. doi: 10.1002/humu.20581. PMID 17621639
- [Background] Rosenberg C, Knijnenburg J, Bakker E, Vianna-Morgante AM, Sloos W, Otto PA, Kriek M, Hansson K, Krepischi-Santos AC, Fiegler H, Carter NP, Bijlsma EK, van Haeringen A, Szuhai K, Tanke HJ. Array-CGH detection of micro rearrangements in mentally retarded individuals: clinical significance of imbalances present both in affected children and normal parents. J Med Genet. 2006 Feb;43(2):180-6. doi: 10.1136/jmg.2005.032268. Epub 2005 Jun 24. PMID 15980116
- [Background] Stankiewicz P, Beaudet AL. Use of array CGH in the evaluation of dysmorphology, malformations, developmental delay, and idiopathic mental retardation. Curr Opin Genet Dev. 2007 Jun;17(3):182-92. doi: 10.1016/j.gde.2007.04.009. Epub 2007 Apr 30. PMID 17467974
- [Background] Zung A, Rienstein S, Rosensaft J, Aviram-Goldring A, Zadik Z. Proximal 19q trisomy: a new syndrome of morbid obesity and mental retardation. Horm Res. 2007;67(3):105-10. doi: 10.1159/000096419. Epub 2006 Oct 19. PMID 17057406